CLINICAL TRIAL: NCT00510497
Title: Phase I/II Evaluation of Therapeutic Immunization With Autologous Dendritic Cells Pulsed With Autologous, Inactivated HIV-1 Infected, Apoptotic Cells
Brief Title: Autologous Dendritic Cell Vaccine in HIV1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sharon Riddler (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Riddler, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Riddler 055794; 5U19AI055794 (NIH)
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections
Keywords: dendritic cell; therapeutic vaccine; HIV-1; apoptotic cells; Phase I/II
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous HIV-1 ApB DC Vaccine (Experimental): Subjects who will receive ApB Dendritic cell vaccine
  Interventions: Biological: Autologous HIV-1 ApB DC Vaccine

INTERVENTIONS:
Biological: Autologous HIV-1 ApB DC Vaccine — Autologous dendritic cells pulsed with autologous, inactivated HIV-1 infected, apoptotic cells given subcutaneously 3 times every other week plus a booster dose 2 weeks after start of treatment interruption

SUMMARY:
This study aims to look at the safety and tolerability of immunization with dendritic cell vaccine prepared using the patient's own cells and virus. It also aims to explore the virologic efficacy of the vaccine as determined by a decrease in the viral load 12 weeks after analytic treatment interruption.

DETAILED DESCRIPTION:
This is a phase I/II, open label, single-arm, single-site clinical trial designed to evaluate the safety and antiviral activity of the ApB DC vaccine, a therapeutic vaccine derived from autologous dendritic cells loaded with autologous HIV-1 infected apoptotic cells. The study will be conducted in three phases. The first is the pre-vaccination phase that includes study entry, isolation of autologous virus, and initiation of antiretroviral therapy. Once the patient's viral load has been suppressed to undetectable levels (<50 copies/mL) and sufficient virus has been isolated, the second phase will begin. This includes leukapheresis in order to harvest monocytes and lymphocytes necessary for vaccine preparation. Three vaccine doses will be administered subcutaneously every other week. Six weeks after the last vaccination, the third phase, analytic treatment interruption (ATI) phase, will begin. A fourth, booster dose of vaccine will be given two weeks after the start of treatment interruption. The treatment interruption will be continued for twelve weeks after which the primary HIV provider will decide whether or not antiretroviral therapy should be restarted. CD4 and viral load will be closely monitored throughout the study especially during treatment interruption. Follow-up will be continued for 24 weeks after the 12-week treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection.
* CD4 greater than or equal to 350 cells/mL within 8 weeks prior to study entry.
* Plasma HIV-1 RNA level of 5000-100,000 copies/mL within 8 weeks prior to study entry.
* Antiretroviral therapy naive.
* Willingness to interrupt ART for at least 12 weeks.
* Written informed consent.

Exclusion Criteria:

* Treatment within 30 days prior to study entry with systemic steroids or other immunosuppressives, or any underlying disease which may require use of such medications during the study period.
* Receipt of any vaccinations other than routine ones within 6 months of study entry
* Pregnancy or breastfeeding
* Previous or current CDC Category C event
* Receipt of any investigational product within 12 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Riddler, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Macatangay BJ, Riddler SA, Wheeler ND, Spindler J, Lawani M, Hong F, Buffo MJ, Whiteside TL, Kearney MF, Mellors JW, Rinaldo CR. Therapeutic Vaccination With Dendritic Cells Loaded With Autologous HIV Type 1-Infected Apoptotic Cells. J Infect Dis. 2016 May 1;213(9):1400-9. doi: 10.1093/infdis/jiv582. Epub 2015 Dec 8. PMID 26647281
- [Result] Whiteside TL, Piazza P, Reiter A, Stanson J, Connolly NC, Rinaldo CR Jr, Riddler SA. Production of a dendritic cell-based vaccine containing inactivated autologous virus for therapy of patients with chronic human immunodeficiency virus type 1 infection. Clin Vaccine Immunol. 2009 Feb;16(2):233-40. doi: 10.1128/CVI.00066-08. Epub 2008 Nov 26. PMID 19038780

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous HIV-1 ApB DC Vaccine
Started | 11
Completed | 8
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 11 particpants were enrolled but one received no study vaccines and was withdrawn and not included in any analyses.
Arm/Group | Autologous HIV-1 ApB DC Vaccine
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 37.9 [20 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Autologous HIV-1 ApB DC Vaccine.
Description: AE graded by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, version 1.0, December 2004
Time Frame: 80 weeks
Measure: Number; unit: participants with Grade 3 events related
Arm/Group | Autologous HIV-1 ApB DC Vaccine
Number analyzed (Participants) | 10
participants with Grade 3 events related | 2

2. Secondary Outcome: Virologic Efficacy (HIV-1 Viral Load at End of ATI Minus Viral Load Prior to ART)
Description: Log10 Change in HIV RNA set point comparing pre-ART to 12 weeks after treatment interruption
Time Frame: at the end of 12 weeks treatment interruption
Measure: Median (Full Range); unit: log10 HIV RNA
Arm/Group | Autologous HIV-1 ApB DC Vaccine
Number analyzed (Participants) | 10
log10 HIV RNA | -0.21 [-0.60 to 0.22]

ADVERSE EVENTS:
Groups:
- Autologous HIV-1 ApB DC Vaccine: Subjects who will receive ApB Dendritic cell vaccine (does not include one enrolled participant who received no study treatment)
  Autologous HIV-1 ApB DC Vaccine: Autologous dendritic cells pulsed with autologous, inactivated HIV-1 infected, apoptotic cells given subcutaneously 3 times every other week plus a booster dose 2 weeks after start of treatment interruption
Arm/Group | Autologous HIV-1 ApB DC Vaccine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous HIV-1 ApB DC Vaccine (N=10)
grade 3 severe pruritus and injection site pain (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days